CLINICAL TRIAL: NCT04511260
Title: Evaluation of the Safety and Efficacy of the NuEra Tight VRF for the Treatment of Vaginal and Vulvar Tissue Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU- NuEra VRF 20-01
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Vagina Atrophy

STUDY DESIGN:
Intervention Model Description: The NuEra device family is FDA cleared (K151296) for a wide range of indications including, but not limited to, selected medical conditions such as temporary relief of pain, muscle spasms, and increase in local circulation. The NuEra Tight - model VRF with the small area handpiece is CE marked in Europe and currently under review by the FDA. In this study, the Radio Frequency treatment will be administered in a continuous motion to the vaginal mucosa and the introitus using the small area handpiece.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VRF Treatment (Experimental): A treatment of the vaginal canal using the NuEra Tight VRF small area handpiece. A treatment of the introitus and vestibule using the NuEra Tight VRF small area hand piece (optional).
  Following screening visit, eligible subjects will be enrolled into the study. Each subject will receive 3 treatments, 4 weeks apart and 2 Follow Up (FU) visits, at 1, and 3 months following the last treatment.
  Interventions: Device: NuEra Tight VRF Handpiece

INTERVENTIONS:
Device: NuEra Tight VRF Handpiece — The VRF is a Model that belongs to the NuEra Tight RF Family, specific for the treatment of small areas.
  The NuEra is FDA cleared (K151296) for a wide range of indications including but not limited to, selected medical conditions such as temporary relief of pain, muscle spasms, and increase in local circulation. The NuEra Tight VRF with the small area handpiece is CE marked in Europe and currently under review by the FDA. The system and its accessories, are intended to be use for a wide range of indications including, but not limited to:
  · Provide heating for the purpose of elevating tissue temperature for selected medical conditions such as temporary relief of pain, muscle spasms, and increase in local circulation of soft tissue.

SUMMARY:
Up to twenty (20) healthy pre- and post-menopausal women with self-reported vaginal laxity will be enrolled in the study.

DETAILED DESCRIPTION:
The treatment will include: A treatment of the vaginal canal using the NuEra Tight VRF small area handpiece. A treatment of the introitus and vestibule using the NuEra Tight VRF small area hand piece (optional).

This is a single center, prospective, open label, single arm study. Following screening visit, eligible subjects will be enrolled into the study. Each subject will receive 3 treatments, 4 weeks apart and 2 Follow Up (FU) visits, at 1, and 3 months following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women age between 35 to 60
* Last vaginal delivery is at least 12 months prior to enrollment
* Self-reported vaginal laxity defined as "very loose," "moderately loose," or "slightly loose" on the Vaginal Laxity Questionnaire (VLQ)
* Sexual activity≥ once per month, with a same partner
* Willing to use contraception for the duration of the study
* Negative urine analysis
* Negative pregnancy test
* Patient is not pregnant nor planning to become pregnant throughout the duration of the study
* Willing to improve vaginal lips / genitals appearance (optional)
* Normal gynecological exam from the recent year
* If taking probiotics and/or any other supplement or suppository as part of daily regimen, willing to maintain same regimen throughout the entire duration of the study
* Able and willing to comply with the treatment/follow-up schedule and requirements ·
* Willing to sign an informed consent

Exclusion Criteria:

* Previous pelvic floor reconstructive surgery with mesh.
* Pelvic organ prolapse (POP) >II according to the pelvic organ prolapse quantification system
* Pregnant or lactating
* Women in post-menopausal stage for more than five years.
* Active genital infection or sexually transmitted diseases
* Subject presenting abnormal Pap smear result from the last five years with any of the following findings according to the Bethesda System (2001) classification: A.. Atypical Squamous Cells-cannot exclude high grade squamous intraepithelial lesion B. Atypical Glandular Cells (Endocervical, Endometrial not otherwise specified) C. High Grade squamous intraepithelial lesion (HSIL)D. Carcinoma
* Patients with implantable devices, such as but not limited to pacemakers, implanted defibrillators, and Cochlear ear implant
* Serious systemic disease or any chronic condition that could interfere with study compliance
* Has metal implant(s) within the treated area, such as surgical clips, plates and screws, intrauterine device (IUD) or artificial joints
* History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of vaginal tissue disease in the treatment area
* Taken part in a clinical trial involving an investigational drug or device within 30 days prior to screening and through the study duration
* Presence of Vulvar lesions or any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety
* Nerve insensitivity to heat anywhere in the treatment area, since ongoing feedback by a patient during a procedure is required
* Previous treatment with a vaginal energy based device, including laser treatment.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of the NuEra small area handpiece | 12 months
  Evaluation of safety and short-term performance of the NuEra small area handpiece treatment on vaginal tissue laxity in pre- and post-menopausal women.
  Change in vaginal laxity as measured by the subject reported laxity rating on a Vaginal Laxity Questionnaire (VLQ) 7-point scale at 1-month follow-up visit compared to baseline. Safety endpoints will include adverse events (AEs) and serious adverse events (SAEs) occurring at any time during the trial or follow-up.

SECONDARY OUTCOMES:
To evaluate the long-term effect on vaginal tissue laxity in pre- and post-menopausal women. | 12 months
  Change in vaginal laxity as measured by the subject reported laxity rating on a Vaginal Laxity Questionnaire (VLQ) 7-point scale at 3-months follow-up visit compared to baseline.
To evaluate the treatment effect on sexual function and overall satisfaction with sexual life | 12 months
  Change in sexual function as evaluated by the subject Female Sexual Function Index (FSFI) at 1, and 3 months follow up visits compared to baseline.
Secondary Objective - 3 | 12 months
  To evaluate improvement in the appearance of the vulva and vaginal lips /genitals (optional)
To evaluate overall improvement following the treatment. | 12 months
  (Optional) Improvement in visual appearance of the vaginal lips /genitals, self-assessed by women at 3 months follow up visit compared to baseline (optional- will be assessed in women receiving treatment for this purpose) - by B&A photos
To evaluate the treatment effect on the general vaginal health. | 12 months
  Subject satisfaction with the treatment using a 5-point Likert scale from post first treatment and after the three months follow up visits by SSQ and Patient Global Impression of Improvement (PGI-I) determined as score of 1-3 (very much better-a little better).
  Change in a physician-reported general vaginal health rating on a VHIS at 1 and 3 months follow up visits compared to baseline.
To evaluate procedure-related subject treatment pain and discomfort | 12 months
  Subject assessment of pain and discomfort that is procedure related using a visual a Pain Visual Analogue Scale (PVAS), evaluated at each treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- NYDerm, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No